CLINICAL TRIAL: NCT00614263
Title: A Prospective, Blinded Study Examining Sedation Levels During Outpatient Colonoscopies
Brief Title: A Study to Examine Levels of Sedation During Outpatient Colonoscopies
Status: Completed | Type: Observational
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 006-005
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Outpatient Colonoscopy
Keywords: Colonoscopy; Sedation levels

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Blinded Group: SEDline output is unknown to anesthesiologist.
- Unblinded Group: SEDline output is known to anesthesiologist.

SUMMARY:
Examine levels of sedation required for patients to comfortably undergo colonoscopy using propofol and if adjunct monitoring equipment promotes patient safety.

DETAILED DESCRIPTION:
Propofol for sedation during outpatient endoscopy has become a popular technique in place of midazolam and opioid sedation. It has been associated with improved patient satisfaction and a faster recovery with less nausea and vomiting. However, there are a number of potential adverse effects associated with propofol. It has no analgesic effects; therefore, when used for moderate sedation procedures it frequently has to provide deeper levels of sedation to allow a painful procedure to be performed.

Some patients are sedated to the level of general anesthesia and may develop respiratory depression or airway obstruction requiring immediate airway support.

We examined the level of sedation required for patients to comfortably undergo routine colonoscopy using propofol and what monitoring system would best predict the patients who might need an airway intervention.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years of age
* ASA classification of I, II, or III

Exclusion Criteria:

* Anesthesiologist plans to use a combination of medications other than propofol for sedation.
* ASA classification IV or higher
* Lesions on forehead or earlobes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient GI clinic
Enrollment: 100 (Actual)
Dates: Start 2006-03; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Examine possible relationships (correlations) between sedation using the SEDLine monitors and level of sedation using the Ramsay Sedation Scale and examine the number and type of airway interventions and clinical signs performed during the procedure. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Ramsay, MD, Principal Investigator — Baylor Research Institute
Locations (1):
- Baylor University Medical Center - Department of Anesthesiology, Dallas, Texas, United States